CLINICAL TRIAL: NCT03020108
Title: The Relation Between Serum Caspase 3, Annexin a2 and Soluble Fas Levels and Severity of Endometriosis
Brief Title: Serum Caspase 3, Annexin a2 and Soluble Fas Levels and Endometriosis
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016/190
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Endometriosis; Apoptotic Pathway Deregulation
MeSH Terms: conditions — Endometriosis | interventions — Blood Specimen Collection; Annexin A2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: The group 1 will comprise of 30 patients with benign ovarian cysts such as mature teratoma or simple serous cysts on ultrasound examination.
  Interventions: Other: Blood sample
- Group 2: The group 2 will comprise of 30 patients with diagnosis of stage 1-2 endometriosis in guidance with the revised American Society for Reproductive Medicine classification.
  Interventions: Other: Blood sample
- Group 3: The group 3 will comprise of 30 patients with diagnosis of stage 3-4 endometriosis in guidance with the revised American Society for Reproductive Medicine classification.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — 2 cc blood samples will be drawn from antecubital vein
  Other Names: Serum caspase 3, annexin a2 and soluble fas levels

SUMMARY:
The study population will comprise of 90 women age varying between 15-55 years, those are candidate for laparoscopic surgery due to definition of >4 cm endometrioma or any other benign ovarian cysts such as mature teratoma or simple serous cysts on ultrasound examination, chronic pelvic pain, infertility. The blood samples will be drawn for analysis of serum biomarkers.

DETAILED DESCRIPTION:
The participants will be accepted for the study between 1st of August 2016 to 30th June 2017. 2 cc blood samples will be drawn from the antecubital vein for serum analysis of caspase 3, annexin a2 and soluble fas levels before the operations. The patients will divide into three groups. The group 1 will comprise of 30 patients with benign ovarian cysts such as mature teratoma or simple serous cysts on ultrasound examination. The group 2 will comprise of 30 patients with diagnosis of stage 1-2 endometriosis in guidance with the revised American Society for Reproductive Medicine classification. The group 3 will comprise of 30 patients with diagnosis of stage 3-4 endometriosis in guidance with the revised American Society for Reproductive Medicine classification. The blood samples will be kept in -80 C degree after centrifuge till at the end of the study.The relation between serum caspase 3, annexin a2 and soluble fas levels and severity of endometriosis will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* The women ages varying between 15-55 years, those are candidate for laparoscopic surgery due to definition of >4 cm endometrioma or any other benign ovarian cysts such as mature teratoma or simple serous cysts on ultrasound examination, chronic pelvic pain, infertility.

Exclusion Criteria:

* The women with malignant diseases, chronic bowel disease, other defined cause of infertility.

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will comprise of women age varying between 15-55 years, those are candidate for laparoscopic surgery due to definition of >4 cm endometrioma or any other benign ovarian cysts such as mature teratoma or simple serous cysts on ultrasound examination, chronic pelvic pain, infertility.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
To determine endometriosis severity with serum markers | 1 year

SECONDARY OUTCOMES:
To determine rectal involvement with serum markers | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Kaya, M.D., Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr Sadi Konuk Teaching and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
To be shared with other researchers after all the data is available

REFERENCES:
- [Background] Flood B, Oficjalska K, Laukens D, Fay J, O'Grady A, Caiazza F, Heetun Z, Mills KH, Sheahan K, Ryan EJ, Doherty GA, Kay E, Creagh EM. Altered expression of caspases-4 and -5 during inflammatory bowel disease and colorectal cancer: Diagnostic and therapeutic potential. Clin Exp Immunol. 2015 Jul;181(1):39-50. doi: 10.1111/cei.12617. Epub 2015 May 6. PMID 25943872
- See also: PUBMED — https://www.ncbi.nlm.nih.gov/pubmed/?term=Altered+expression+of+caspases-4+and+-5+during+inflammatory+bowel+disease+and+colorectal+cancer%3A+diagnostic+and+therapeutic+potential